CLINICAL TRIAL: NCT00665145
Title: A Phase 2 Study of Stem-Cell-Mobilization in Subjects With Diabetic Neuropathy Receiving SB-509
Brief Title: Stem Cell Mobilization in Diabetic Neuropathy Subjects Receiving SB-509
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Ely Benaim, M.D., Vice President, Clinical Affairs, Sangamo BioSciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SB-509-0703
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy
Keywords: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy; Stem Cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Cohort 1
  Interventions: Drug: SB-509
- 2 (Experimental): Cohort 2
  Interventions: Drug: SB-509
- 3 (Placebo Comparator): Cohort 3
  Interventions: Drug: Placebo
- 4 (Experimental): Cohort 4
  Interventions: Drug: SB-509

INTERVENTIONS:
Drug: SB-509 — Active drug
  Arms: 1
Drug: SB-509 — Active drug
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3
Drug: SB-509 — Active drug
  Arms: 4

SUMMARY:
The primary and secondary objectives of this study are:

Primary: To evaluate stem-cell-mobilization in subjects with diabetic neuropathy receiving SB-509. Stem cell mobilization will be assessed by evaluating the presence of stem cells circulating in peripheral blood.

Secondary: To evaluate the safety of SB-509 in subjects treated with SB-509 with diabetic neuropathy; and to compare the effect of SB-509 versus placebo on a pre-defined multi-endpoint analysis that includes visual analog scale for pain intensity (VASPI), total neuropathy score (TNS), evoked nerve conduction velocity (NCV) and quantitative sensory testing (QST)

DETAILED DESCRIPTION:
SB-509 contains the gene (DNA-a kind of biological "blueprint") for a protein. When a researcher injects SB-509 into your legs, the drug enters the muscle and nerve cells around the injection site and causes these cells to make a protein. This protein causes your cells to increase production of another protein called vascular endothelial growth factor (VEGF), which may improve the structure and function of nerves. In addition, there are changes in the levels of 28 additional proteins in your cells. These proteins function to promote the growth of cells, are structures in cells, help synthesize products, and affect immune cells, and some have unknown functions. This increase in your own VEGF proteins may protect and repair the damaged nerves caused by diabetic neuropathy.

This study is intended to further evaluate the mechanism of SB-509 action.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

* Have a clinical diagnosis of diabetes mellitus type I or II for at least 12 months prior to the study.
* Have received a diagnosis of sensorimotor diabetic neuropathy from a neurologist (a doctor who specializes in disorders of the nervous system) or endocrinologist (a doctor who specializes in diabetes).
* Have reduced nerve conduction velocity in any lower extremity nerve: peroneal, tibial or sural due to diabetic polyneuropathy
* If female and of childbearing potential, agree to use a medically acceptable physical barrier method during the study.
* Have blood pressure < 140/90 mm Hg
* Body mass index (BMI) < 38 kg/m2

Key Exclusion Criteria:

Subjects with the following are NOT eligible to participate in this study:

* Have moderate to severe ischemic heart disease, any history of congestive heart failure, or have had a myocardial infarction (heart attack) within the previous 6 months.
* Have chronic foot or leg ulcers for >1 month, gangrene in the legs, or any previous amputation of the lower extremity.
* Have a history of cancer within the past 5 years (except for curable non-melanoma cancer of the skin, superficial bladder cancer in complete remission, or any other cancer that has been in complete remission for at least 5 years).
* Have colon polyps. If patients have a history of benign colonic polyps that have been removed, they must have evidence of a normal colonoscopy within the last 12 months.
* Require any drug that depresses patients' immune systems (such as methotrexate, cyclophosphamide, or cyclosporine) when they receive the study drug and for 30 days afterwards.
* Have a known disorder that affects patients' immune systems (such as HIV/AIDS, hepatitis B virus [HBV], hepatitis C virus [HCV], sarcoidosis, tuberculosis, rheumatoid arthritis, or autoimmune disorders).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Stem cells circulating in peripheral blood | One year

SECONDARY OUTCOMES:
Safety and Efficacy of SB-509 | One year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - La Jolla, California
  - Walnut Creek, California
  - Houston, Texas
  - San Antonio, Texas

REFERENCES:
- See also: Company website — http://www.sangamo.com